CLINICAL TRIAL: NCT02992132
Title: A Double-Blind, Placebo-Controlled Study to Examine the Safety and Efficacy of Pimavanserin for the Treatment of Agitation and Aggression in Alzheimer's Disease
Brief Title: Study to Examine the Safety and Efficacy of Pimavanserin for the Treatment of Agitation and Aggression in Alzheimer's Disease (SERENE)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACP-103-032; 2016-001127-32 (EudraCT Number)
Record Dates: First submitted 2016-12-12; First posted 2016-12-14 (Estimated); Results first posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Agitation and Aggression in Alzheimer's Disease
MeSH Terms: conditions — Psychomotor Agitation | interventions — pimavanserin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pimavanserin 34 mg (Experimental): Drug- pimavanserin tartrate, 34 mg, taken as two 17 mg tablets, once daily by mouth
  Interventions: Drug: Pimavanserin 34 mg
- Pimavanserin 20 mg (Experimental): Drug- pimavanserin tartrate, 20 mg, taken as two 10 mg tablets, once daily by mouth
  Interventions: Drug: Pimavanserin 20 mg
- Placebo (Placebo Comparator): Placebo, taken as two tablets, once daily by mouth
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pimavanserin 34 mg — Pimavanserin 34 mg, tablet, taken as two 17 mg tablets, once daily by mouth
  Arms: Pimavanserin 34 mg
Drug: Pimavanserin 20 mg — Pimavanserin 20 mg, tablet, taken as two 10 mg tablets, once daily by mouth
  Arms: Pimavanserin 20 mg
Other: Placebo — Placebo, taken as two tablets, once daily by mouth
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of pimavanserin compared with placebo in treatment of agitation and aggression after 12 weeks of treatment

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 50 years of age or older
2. Can understand the nature of the trial and protocol requirements and provide signed informed consent

   * from patient, if deemed competent to provide consent
   * from an appropriate person (e.g. patient's Legally Authorized Representative (LAR) with the patient's assent) if patient is deemed not competent to provide informed consent.
3. Has a diagnosis of probable AD according to the National Institute on Aging-Alzheimer's Association (NIA-AA) guidelines
4. Meets criteria for agitation according to the International Psychogeriatric Association (IPA) guidelines
5. Lives at home or in an assisted living or care facility (but has the capacity to visit the clinic as an outpatient). Subjects must have been at their current location for at least 3 weeks prior to Screening and plan to remain at the same location for the duration of the trial.
6. Has a designated study partner/caregiver who is in contact with the patient at least 3 times a week on 3 separate days
7. Female patients must be of non-childbearing potential or must agree to use an acceptable method of contraception or abstinence , for at least 1 month prior to randomization, during the study, and 1 month following completion of the study
8. The patient and caregiver are willing and able to participate in all schedule evaluations and complete all required tests

Exclusion Criteria:

1. The agitation/aggression is attributable to concomitant medications, environmental conditions, substance abuse, or active medical or psychiatric condition
2. Patient is receiving skilled nursing care for any medical condition other than dementia
3. Treatment with an antipsychotic medication within 2 weeks of Baseline visit or 5 half lives, whichever is longer
4. Patient or study partner/caregiver has a medical condition (e.g., hearing, vision impairments) that would impair the ability to perform the study assessments.
5. Has had a myocardial infarction within the last six months
6. Has a history or symptoms of long QT syndrome
7. Has a history of a significant psychotic disorder before or during the diagnosis of probable Alzheimer's disease (including, but not limited to schizophrenia or bipolar disorder)
8. Patient is bedridden or has any significant medical condition that is unstable and would place the patient at undue risk from study drug or study procedures 9. Has a sensitivity to pimavanserin or its excipients

10. Has previously participated in a clinical study with pimavanserin

11. Has a Global Clinician Assessment of Suicidality (GCAS) score of 3 or 4 based on Investigator's assessment of behavior within the last 3 months at Screening or since last visit at Baseline

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2016-11; Primary Completion 2018-01-25 (Actual); Study Completion 2018-02-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (55):
- United States (33):
  - Costa Mesa, California
  - Fresno, California
  - Fullerton, California
  - Los Angeles, California
  - Pasadena, California
  - San Diego, California
  - Danbury, Connecticut
  - Washington D.C., District of Columbia
  - Boca Raton, Florida
  - Deerfield Beach, Florida
  - Miami, Florida
  - Naples, Florida
  - Atlanta, Georgia
  - Bangor, Maine
  - Quincy, Massachusetts
  - Clinton Township, Michigan
  - Flowood, Mississippi
  - Jackson, Mississippi
  - Eatontown, New Jersey
  - Marlton, New Jersey
  - Toms River, New Jersey
  - Albuquerque, New Mexico
  - Charlotte, North Carolina
  - Oklahoma City, Oklahoma
  - Medford, Oregon
  - Jenkintown, Pennsylvania
  - Norristown, Pennsylvania
  - Willow Grove, Pennsylvania
  - Charleston, South Carolina
  - Nashville, Tennessee
  - DeSoto, Texas
  - Salt Lake City, Utah
  - Spokane, Washington
- Chile (3):
  - Valdivia, Los Ríos Region
  - Antofagasta
  - Santiago
- France (5):
  - Toulouse, Cedex 9
  - Paris
  - Saint-Herblain
  - Strasbourg
  - Villeurbanne
- Spain (9):
  - Algorta, Vizcaya
  - Córdoba
  - Elche
  - Madrid
  - Palma de Mallorca
  - Pamplona
  - Santa Coloma de Gramenet
  - Terrassa
  - Zaragoza
- United Kingdom (5):
  - Swindon, Wiltshire
  - Bath
  - Isleworth
  - Manchester
  - Northampton

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was planned to be conducted in approximately 432 subjects. For business reasons, and not related to safety, recruitment of subjects was stopped after 111 subjects were randomized. The last subject was randomized on 2 Nov 2017.
Pre-assignment Details: The screening visit was followed by a 2- to 4-week screening period, including wash-out of antipsychotic agents which were prohibited during the Treatment period (exception: protocol specified agents). Subjects had to be on stable doses of permitted medications for >=4 weeks before Baseline (>=12 weeks for cholinesterase inhibitors and memantine).
Period: Overall Study
Arm/Group | Placebo | Pimavanserin 20 mg | Pimavanserin 34 mg
Started | 40 | 35 | 36
Completed | 27 | 27 | 29
Not Completed | 13 | 8 | 7
Not completed — Adverse Event | 4 | 1 | 3
Not completed — Lack of Efficacy | 2 | 0 | 0
Not completed — Non-compliance with study drug | 2 | 0 | 0
Not completed — Progressive disease | 1 | 0 | 0
Not completed — Protocol Violation | 2 | 2 | 0
Not completed — Caregiver withdrew consent | 2 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 2 | 1
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All patients randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pimavanserin 20 mg | Pimavanserin 34 mg | Total
Number analyzed (Participants) | 40 | 35 | 36 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.9 (7.58) | 76.5 (8.74) | 75.0 (7.90) | 76.8 (8.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 15 | 18 | 58
  Male | 15 | 20 | 18 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 16 | 17 | 53
  Not Hispanic or Latino | 17 | 15 | 18 | 50
  Unknown or Not Reported | 3 | 4 | 1 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 36 | 31 | 32 | 99
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Cohen-Mansfield Agitation Inventory (CMAI)
Description: The Cohen-Mansfield Agitation Inventory (CMAI) is a 29-item scale to assess agitation. Each item is rated on a 7-point scale of frequency, from least (1) to most frequent (7). Items are summed to calculate the CMAI total score. The CMAI total score has a range of 29-203 points; higher scores indicate more severe agitation
Time Frame: Baseline to 12 weeks
Population: Full Analysis set, i.e. patients who had been randomized and treated and had both a baseline value and at least 1 post-baseline value for the CMAI total score.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Pimavanserin 20 mg | Pimavanserin 34 mg
Number analyzed (Participants) | 37 | 34 | 35
score on a scale
  Baseline | 70.3 (4.5) | 56.9 (2.2) | 68.0 (3.3)
  Week 12: number analyzed (Participants) | 29 | 28 | 29
  Week 12 | 54.3 (4.3) | 52.5 (4.3) | 53.7 (3.0)
  Week 12 change from baseline: number analyzed (Participants) | 29 | 28 | 29
  Week 12 change from baseline | -16.8 (5.0) | -3.7 (3.7) | -12.3 (2.7)
Statistical Analysis 1: Comparison: Placebo vs Pimavanserin 20 mg; Mixed-effect model repeated measures (MMRM), with the dependent variable being the change from Baseline in CMAI total score; Test type: Superiority; Difference in LSM = 5.1, 95% CI 2-sided [-4.8 to 15.0], Standard Error of Mean 5.0
Statistical Analysis 2: Comparison: Placebo vs Pimavanserin 34 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Difference in LSM = 1.0, 95% CI 2-sided [-8.5 to 10.5], Standard Error of Mean 4.8

2. Secondary Outcome: Zarit Burden Interview
Description: The Zarit Burden Interview (ZBI) assess the stresses experienced by caregivers of patients with dementia. It assesses 22 questions about the impact of the patient's disabilities on the caregiver's life, each rated from least (0) to most (4) frequent. Items are summed to calculate the ZBI total score. The ZBI total score ranges from 0 to 88; higher scores denoting more stresses experienced by caregivers.
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Pimavanserin 20 mg | Pimavanserin 34 mg
Number analyzed (Participants) | 34 | 33 | 32
score on a scale
  Baseline | 41.5 (2.6) | 40.8 (2.4) | 41.7 (2.5)
  Week 12: number analyzed (Participants) | 28 | 27 | 27
  Week 12 | 37.0 (3.2) | 36.8 (3.7) | 35.7 (3.5)
  Week 12 change from baseline: number analyzed (Participants) | 28 | 27 | 27
  Week 12 change from baseline | -6.5 (2.3) | -4.9 (2.3) | -5.5 (2.5)

ADVERSE EVENTS:
Time Frame: From the time of informed consent through the completion of procedures at the Week 12 visit (for subjects continuing into an Open-Label Extension study) or through to 30 days after the last dose of study drug (for all other subjects)
Arm/Group | Placebo | Pimavanserin 20 mg | Pimavanserin 34 mg
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/35 | 0/36
Serious Adverse Events (participants affected / at risk) | 3/40 | 4/35 | 3/36
Other Adverse Events (participants affected / at risk) | 11/40 | 15/35 | 15/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=40) | Pimavanserin 20 mg (N=35) | Pimavanserin 34 mg (N=36)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=40) | Pimavanserin 20 mg (N=35) | Pimavanserin 34 mg (N=36)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (2) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2)
Agitation (Psychiatric disorders) | 5 (5) | 5 (5) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 4 (5) | 3 (3)

LIMITATIONS AND CAVEATS:
The original study (n=432) was powered to detect a treatment effect on CMAI, however recruitment was discontinued early for business reasons and amended accordingly The final study (n=111) was no longer adequately powered to detect a treatment effect

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish the study results, relative to his/her own patients, only after review, comment and approval by the sponsor. No publication of confidential information shall be made without the sponsor's prior written consent. At least 60 days prior to submitting a manuscript or prior to any public presentation, a copy of the manuscript or presentation will be provided to the sponsor for review and comment. The sponsor has 60 days to review and comment.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-11-22): https://cdn.clinicaltrials.gov/large-docs/32/NCT02992132/SAP_000.pdf
  • Study Protocol (2017-12-28): https://cdn.clinicaltrials.gov/large-docs/32/NCT02992132/Prot_001.pdf